CLINICAL TRIAL: NCT03503084
Title: The Effect of Tai Chi Chuan on the Endothelin, Insulin, Blood Lipid, Blood Sugar, Aldosterone and Hemodynamics in the Elderly Adults
Brief Title: Short-term Effects of Tai Chi Chuan Exercise on the Regulation of Lipid and Glucose Metabolisms and Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Cheng-Deng Kuo, Principal Investigator, Changhua Christian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: V98E2-014
Record Dates: First submitted 2018-03-30; First posted 2018-04-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Physiological Effect of TCC on Glucose Metabolism
Keywords: Tai Chi Chuan; insulin resistance; cholesterol; endothelin-1
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Twenty-one TCC practitioners and nineteen normal controls were included in this study. The hemodynamics, serum insulin, indices of insulin resistance/sensitivity, serum endothelin-1 (ET-1), blood lipids and aldosterone before and 30 min after a rest or a session of classical Yang's TCC exercise were compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCC group (Experimental): Classical Yang's TCC exercise
  Interventions: Behavioral: Classical Yang's TCC exercise

INTERVENTIONS:
Behavioral: Classical Yang's TCC exercise

SUMMARY:
The short term effects of TCC exercise are the significant increase in serum insulin and insulin resistance, and the significant decrease in serum TC, HDL-C, ET-1 and insulin sensitivity in TCC practitioners. TCC might be benefit the health of its practitioners through the regulation of lipid and glucose metabolism and endothelial function.

DETAILED DESCRIPTION:
Tai Chi Chuan (TCC) has been shown to be beneficial to the health. However, its effects on lipid and glucose metabolism are not fully understood. This study investigated the short term effect of TCC exercise on lipid and glucose metabolism and endothelial function in TCC practitioners. Twenty-one TCC practitioners and nineteen normal controls were included in this study. The hemodynamics, serum insulin, indices of insulin resistance/sensitivity, serum endothelin-1 (ET-1), blood lipids and aldosterone before and 30 min after a rest or a session of classical Yang's TCC exercise were compared.

ELIGIBILITY:
Inclusion Criteria:

* TCC practitioners in a TCC training center in Taiwan over 50 years of age
* Healthy subjects without TCC experience over 50 years of age

Exclusion Criteria:

* Subjects who had major cardiopulmonary disease
* Subjects who have diabetes mellitus, renal or liver disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
change in quantitative insulin sensitivity check index | before and 30 minutes after the completion of TCC exercise
  change in insulin sensitivity due to TCC

SECONDARY OUTCOMES:
change in serum total cholesterol | before and 30 minutes after the completion of TCC exercise
  change in serum total cholesterol due to TCC
change in homeostasis model assessment-estimated insulin resistance | before and 30 minutes after the completion of TCC exercise
  change in insulin resistance by TCC

OTHER OUTCOMES:
change in serum triglyceride | before and 30 minutes after the completion of TCC exercise
  change in serum level of triglyceride due to TCC
change in serum low density lipoprotein | before and 30 minutes after the completion of TCC exercise
  change in serum level of low density lipoprotein due to TCC
change in serum high density lipoprotein | before and 30 minutes after the completion of TCC exercise
  change in serum level of high density lipoprotein due to TCC
change in serum insulin | before and 30 minutes after the completion of TCC exercise
  change in serum level of insulin due to TCC
change in serum endothelin-1 | before and 30 minutes after the completion of TCC exercise
  change in serum level of endothelin-1 due to TCC
change in serum aldosterone | before and 30 minutes after the completion of TCC exercise
  change in serum level of aldosterone due to TCC

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Deng Kuo, MD,PhD, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Wan-An Lu, Yilan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) are available after the manuscript has been accepted for publication

REFERENCES:
- [Result] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Result] Muniyappa R, Lee S, Chen H, Quon MJ. Current approaches for assessing insulin sensitivity and resistance in vivo: advantages, limitations, and appropriate usage. Am J Physiol Endocrinol Metab. 2008 Jan;294(1):E15-26. doi: 10.1152/ajpendo.00645.2007. Epub 2007 Oct 23. PMID 17957034
- [Result] Couillard C, Despres JP, Lamarche B, Bergeron J, Gagnon J, Leon AS, Rao DC, Skinner JS, Wilmore JH, Bouchard C. Effects of endurance exercise training on plasma HDL cholesterol levels depend on levels of triglycerides: evidence from men of the Health, Risk Factors, Exercise Training and Genetics (HERITAGE) Family Study. Arterioscler Thromb Vasc Biol. 2001 Jul;21(7):1226-32. doi: 10.1161/hq0701.092137. PMID 11451756
- [Result] Lu WA, Kuo CD. The effect of Tai Chi Chuan on the autonomic nervous modulation in older persons. Med Sci Sports Exerc. 2003 Dec;35(12):1972-6. doi: 10.1249/01.MSS.0000099242.10669.F7. PMID 14652490
- [Result] Lu WA, Kuo CD. Three months of Tai Chi Chuan exercise can reduce serum triglyceride and endothelin-1 in the elderly. Complement Ther Clin Pract. 2013 Nov;19(4):204-8. doi: 10.1016/j.ctcp.2013.06.007. Epub 2013 Jul 27. PMID 24199974
- [Result] Salgado AL, Carvalho Ld, Oliveira AC, Santos VN, Vieira JG, Parise ER. Insulin resistance index (HOMA-IR) in the differentiation of patients with non-alcoholic fatty liver disease and healthy individuals. Arq Gastroenterol. 2010 Apr-Jun;47(2):165-9. doi: 10.1590/s0004-28032010000200009. PMID 20721461
- [Result] Katz A, Nambi SS, Mather K, Baron AD, Follmann DA, Sullivan G, Quon MJ. Quantitative insulin sensitivity check index: a simple, accurate method for assessing insulin sensitivity in humans. J Clin Endocrinol Metab. 2000 Jul;85(7):2402-10. doi: 10.1210/jcem.85.7.6661. PMID 10902785